CLINICAL TRIAL: NCT05879406
Title: A 12-week, Randomized, Double-blind, Placebo Controlled Study Evaluating the Efficacy and Safety of Clear Skin Formula on Mitigating Mild to Moderate Non-cystic Acne in Young Healthy Adults
Brief Title: A Study to Evaluate the Efficacy and Safety of Clear Skin Formula on Mitigating Mild to Moderate Non-cystic Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: Grove Acquisition Subsidiary dba VitaMedica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VM-CSF-01[
Record Dates: First submitted 2023-05-04; First posted 2023-05-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-05

CONDITIONS: Non-Cystic Acne

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled study evaluating the efficacy and safety
Who Masked: Participant, Care Provider
Masking Description: Randomized, double-blind, placebo controlled study evaluating the efficacy and safety
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VitaMedica® Clear Skin Formula capsules (Active Comparator): Storage Instructions: Store in a cool, dry place. Contents: 60 Capsules Directions for Use: As a dietary supplement, take two capsules with food. Caution: Do not take if safety seal on bottle is broken. KEEP OUT OF REACH OF CHILDREN.
  Interventions: Dietary Supplement: VitaMedica® Clear Skin Formula capsules
- Placebo Capsules (Placebo Comparator): Storage Instructions: Store in a cool, dry place. Contents: 60 Capsules Directions for Use: As a dietary supplement, take two capsules with food. Caution: Do not take if safety seal on bottle is broken. KEEP OUT OF REACH OF CHILDREN.
  Interventions: Other: Placebo Capsules

INTERVENTIONS:
Dietary Supplement: VitaMedica® Clear Skin Formula capsules — After an initial screening period to determine eligibility, subjects will be randomly assigned to one of the following treatment arms: VitaMedica® Clear Skin Formula vs. Placebo for the duration of the twelve (12) week trial
  Ingredients:
  Vitamin A (from Betatene® Carotenoid Blend) (7,500 IU/2,250 mcg RAE) Vitamin A (from Retinyl Palmitate) (5,000 IU/1,500 mcg RAE) Vitamin C (as Ascorbic Acid) (60 mg) Vitamin E (from d-alpha-Tocopheryl Acid Succinate) (30 IU/20 mg) Zinc (from Zinc Bisglycinate Chelate) (24 mg) Selenium (from Selenium Glycinate) (48 mcg) Chromium (from Chromium Nicotinate Glycinate Chelate) (150 mcg) MSM (Methylsulfonylmethane) (200 mg) Bromelain (200 mg) Burdock (Arctium lappa) root (50 mg) Oregon Grape (Mahonia aquifolium) root (25 mg) Dandelion (Taraxacum officinale) root (50 mg) Yellow Dock Extract (Rumex crispus) root (50 mg) Hypromellose Microcrystalline cellulose Magnesium Stearate Silicon Dioxide
  Arms: VitaMedica® Clear Skin Formula capsules
Other: Placebo Capsules — After an initial screening period to determine eligibility, subjects will be randomly assigned to one of the following treatment arms: VitaMedica® Clear Skin Formula vs. Placebo for the duration of the twelve (12) week trial
  Ingredients:
  Magnesium Stearate (VEG) (NON-GMO) Silica (As Silicon Dioxide) Micro Cellulose (MCG) (NON-GMO)
  Arms: Placebo Capsules

SUMMARY:
The goal of this clinical trial is to compare Clear Skin Fomula Supplement to Placebo in healthy men and women ages 18-40 to mitigate mild to moderate non-cystic acne over the course of 12 weeks. Participants will be asked to take a daily supplement, have photos of their face taken and answer questionnaires related to their acne.

DETAILED DESCRIPTION:
Non-cystic acne is a common disorder of sebaceous follicles most prevalent among teenagers, has a multifactorial etiology often triggered by the increase in androgen production, and yet, approximately 3% to 8% of adults 25 to 44 years of age continue to have breakouts. The pathogenesis is complex and appears to involve 4 primary features: increased stimulation of sebum gland activity, increased bacterial proliferation (especially Propionibacterium acnes), abnormal follicular hyperkeratinization and resultant obstruction of the sebaceous follicles, and the release of inflammatory mediators. These changes in non-cystic acne patients result in the formation of non-inflammatory and inflammatory lesions including superficial pustules such as comedones (popularly known as "blackheads" or "whiteheads") and papules. The areas most affected by the non-cystic acne include the pilosebaceous follicles of the head and upper trunk, where the sebaceous glands are particularly active.

With the complexity of the pathogenic mechanisms leading to non-cystic acne, consensus guidelines recommend the use of combination therapy including various topical applications (retinoids, antibiotics, salicylic acid, dapsone); oral medications (antibiotics, oral contraceptives, anti-androgen agents, isotretinoin); and numerous other therapies (light therapy, steroid injection, chemical peel, comedone extraction). While the standard treatments for non-cystic acne have varying degrees of effectiveness, significant side-effects including but not limited to skin dryness, irritation, redness, and disturbance of the skin and gut microbiome can occur. Importantly, overprescribing of antibiotics has contributed to antibiotic resistance and reduction of efficacy for these medications.

Use of nutritional supplements as a component of non-cystic acne treatments has increased in popularity due to credible clinical validation and acceptance by the medical community, as well as reported advantages such as better patient tolerance, minimal side-effects, widespread availability and reduced expense versus prescription and over the counter products. Specifically Vitamin A and Carotenoids (the basis of the prescription Isotretinoin), have shown to serve as substitutes when Isotretinoin is inaccessible. Since the progression of non-cystic acne produces free radicals, oxidative stress may be implicated in the origin of non-cystic acne, so that antioxidant vitamins may be valuable adjuncts in non-cystic acne treatment. Additional Vitamins and Minerals have also shown substantial improvement in non-cystic acne.

Although a clinical study has not been previously conducted on VitaMedica® Clear Skin Formula, extensive clinical and patient use data support further investigation. For two decades hundreds of aesthetic and dermatology medical practices in the U.S. have utilized or recommended this VitaMedica® Clear Skin Formula as a safe and effective adjunctive therapy for their non-cystic acne patients. To date, more than 140,000 individual patients have used this dietary supplement in conjunction with their usual treatment regimens.

As the causes of non-cystic acne are multifactorial, and resources to common prescription medications can be costly and frequently ineffective, finding alternative therapies is crucial. Investigators know that diet and nutrition affect all conditions of the skin, gut and brain, so it is logical to infer that vitamins and supplements, while proving successful in treating a multitude of dermatologic conditions, including hair loss, connective tissue disorders, psoriasis and other papulosquamous disorders, could also help mitigate non-cystic acne. Because of this data, two decades ago the VitaMedica® Clear Skin Formula was developed. It includes the following ingredients:

Vitamin A (from Betatene® Carotenoid Blend) (7,500 IU/2,250 mcg RAE) Vitamin A (from Retinyl Palmitate) (5,000 IU/1,500 mcg RAE) Vitamin C (as Ascorbic Acid) (60 mg) Vitamin E (from d-alpha-Tocopheryl Acid Succinate) (30 IU/20 mg) Zinc (from Zinc Bisglycinate Chelate) (24 mg) Selenium (from Selenium Glycinate) (48 mcg) Chromium (from Chromium Nicotinate Glycinate Chelate) (150 mcg) MSM (Methylsulfonylmethane) (200 mg) Bromelain (200 mg) Burdock (Arctium lappa) root (50 mg) Oregon Grape (Mahonia aquifolium) root (25 mg) Dandelion (Taraxacum officinale) root (50 mg) Yellow Dock Extract (Rumex crispus) root (50 mg) Hypromellose Microcrystalline cellulose Magnesium Stearate Silicon Dioxide

This is a twelve (12) week double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of VitaMedica® Clear Skin Formula in the mitigation of mild to moderate non-cystic acne in young, healthy males and females ages 18-40. After an initial screening period to determine eligibility, subjects will be randomly assigned to one of the following treatment arms: VitaMedica® Clear Skin Formula vs. Placebo for the duration of the twelve (12) week trial at Visit 2 (Day 0). Subjects will return to the study site at Visit 3 (Day 14), Visit 4 (Day 28), Visit 5 (Day 56) and Visit 6 (Day 84) for assessments.

The primary efficacy endpoints are to be evaluated using the following parameters:

1. Change in inflammatory lesion counts from Baseline to Day 84.
2. Change in non-inflammatory lesion counts from Baseline to Day 84.
3. Percentage/Proportion of subjects who achieve at least a one-grade reduction in the Modified IGA Score from Baseline to Day 84.

The secondary efficacy endpoints are to be evaluated using the following parameters:

1. Improvement in Non-Cystic Acne Quality of Life questionnaire scores from Baseline to Day 84.
2. Improvement in Non-Cystic Acne Self Assessment questionnaire scores from Baseline to Day 84.
3. Favorable Analysis of the Clear Skin Formula Supplement Subject Satisfaction questionnaire at Day 84.

The tertiary efficacy endpoints are to be evaluated using the following parameters:

1) Improvement from Baseline to Day 84 in the VISIA photography imaging of the left, right and front views of the face to include the (1) Percentile Rating, (2) Score Rating and (3) Feature Count Rating for Wrinkles, Texture, Pores, Red Areas and Porphyrins.

The tolerability and safety objectives of this study are:

To determine the nature, severity and frequency of the AEs rate and the local cutaneous tolerability of VitaMedica® Clear Skin Formula compared to the placebo.

The tolerability and safety endpoints to be assessed include the following:

1. The frequency of both local and systemic AEs
2. Investigator Tolerability Assessment (erythema, edema, dryness, scaling, hypopigmentation and hyperpigmentation) and Subject Tolerability Self-Assessment (itching, burning and stinging) at Baseline and at all study visits.
3. Changes from baseline to Day 84 in all safety laboratory values as summarized using descriptive statistics by treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or females of all Fitzpatrick Skin Types between 18 and 40 years of age.
2. Subjects must be willing to provide verbal understanding and sign an Informed Consent Form, HIPAA Form and Photography Release Form approved by the Institutional Review Board.
3. Subjects must be in general good health, as determined by the Investigator.
4. Subjects must be willing and able to attend all study visits and comply with the test product daily instructions.
5. Subjects must be willing to have VISIA facial photography imaging of their entire face for overall evaluation of their skin at all Visits.
6. Subjects must be willing and able to complete and understand the various rating questionnaires.
7. Subjects must have a Modifed IGA score of 2 (mild) or 3 (moderate) at the Baseline Visit.
8. Subjects must have a facial non-cystic acne inflammatory lesion (papules and pustules) count with no less than 10 but no more than 50.
9. Subjects must have a facial non-cystic acne non-inflammatory lesion (open and closed comedones) count with no less than 10 but no more than 100.
10. Females of child bearing potential (FOCBP) and females who are premenses must be willing to practice effective contraception for the duration of the study. (Effective contraception is defined as stabilized on oral contraceptive for at least 3 months, intrauterine device, condom with spermicide, diaphragm with spermicide, implant, NuvaRing®, injection, transdermal patch or abstinence.) Females on birth control pills must have taken the same type pill for at least 3 months prior to entering the study and must not change type during the study. Those who have used birth control pills in the past must have discontinued usage at least 3 months prior to the start of the study. Women who use birth control for non-cystic acne control only should be excluded.
11. Premenses females and FOCBP must have a negative urine pregnancy test at the Baseline Visit.
12. Subjects must be willing to comply with study instructions and return to the clinic for required visits.
13. If a cleanser, moisturizer or sunscreen is needed during the study, subjects must be willing to use the cleanser, moisturizer and sunscreen provided by the Sponsor.
14. If the subject wears makeup, they must agree to use non-comedogenic makeup.
15. Male subjects facial area must be clean-shaven for all study visits as to not interfere with study assessment.

Exclusion Criteria:

* Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study. 2. Any dermatological conditions on the face that could interfere with clinical evaluations such as cystic acne, acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, Gram-negative folliculitis, dermatitis, eczema. 3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.

  4. Subjects with more than 50 facial non-cystic acne inflammatory lesions (papules and pustules).

  5. Subjects with more than 100 facial non-cystic acne non-inflammatory lesions (open and closed comedones) 6. Subjects with facial acne cysts. 7. Subjects with a facial beard or mustache that could interfere with the study assessments.

  8. Subject has a history of experiencing significant burning or stinging when applying any facial treatment (eg, makeup, soap, masks, washes, sunscreens, etc) to their face. 9. Female subjects who are pregnant, nursing mothers, planning a pregnancy during the course of the study, or become pregnant during the study. 10. If female, subject has a history of hirsutism, polycystic ovarian disease or clinically significant menstrual irregularities. 11. History of regional enteritis, ulcerative colitis, inflammatory bowel disease, pseudomembranous colitis, chronic or recurrent diarrhea, or antibiotic-associated colitis. 12. Treatment of any type of cancer within the last 6 months, with the exception of complete surgical excision of skin cancer outside the treatment area. 13. Subjects who have not undergone the specified washout period(s) for the following topical preparations/physical treatments used on the face or subjects who require the concurrent use of any of the following in the treatment area:

Topical astringents and abrasives on the face 1 week Non-allowed moisturizers or sunscreens on the face 1 week Non-cystic Acne surgery 1 week Antibiotics on the face 2 weeks Other topical non-cystic acne drugs on the face 2 weeks Soaps containing antimicrobials on the face 2 weeks Light (e.g. LED, PDT) therapy on the face 2 weeks Anti-inflammatory agents and corticosteroids on the face 4 weeks Retinoids, including retinol on the face 4 weeks Chemical peel/Microdermabrasion on the face 4 weeks Laser therapy on the face 4 weeks

14. Subjects who have not undergone the specified washout period(s) for the following systemic medications or subjects who require the concurrent use of any of the following systemic medications:

High Dose Vitamin A and Beta-carotene Supplements 2 weeks Corticosteroids (including intramuscular injections) (inhaled corticosteroids are allowed) 4 weeks Antibiotics 4 weeks Other systemic treatments 4 weeks Systemic retinoids 6 months

15. Subject intends to use a tanning booth or sunbathe during the study. 16. Subjects who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function. 17. Subjects with any underlying disease that the investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | Baseline to Day 84
  Papule - A small, solid elevation less than 5 mm in diameter. Most of the lesion is above the surface of the skin.
  Pustule - A small circumscribed elevation less than 5 mm in diameter that contains yellow-white exudate.
Change in non-inflammatory lesion counts | Baseline to Day 84
  Open Comedone - (Blackhead) A lesion in which the follicle opening is widely dilated with the contents protruding out onto the surface of the skin, with exposed keratin cells giving the plug a black appearance.
  Closed Comedone - (Whitehead) A lesion in which the follicle opening is closed, with sebum buildup, which in turn cause the skin around the follicle to thin and become elevated with a white appearance.
Percentage/Proportion of subjects who achieve at least a one-grade reduction in the Modified IGA Score | Baseline to Day 84
  Modified Investigator Global Assessment (IGA) Scale for Non-Cystic Acne The Investigator will use the Modified Investigator Global Assessment (IGA) Scale to assess the severity of a subjects' non-cystic acne. The Modified IGA Scale is a static evaluation of global severity representing clinically meaningful graduations of non-cystic acne. The Modified IGA should be performed prior to the lesion count. The Modified IGA will be performed at visits: Baseline, Day 14, Day 28, Day 56,Day 84 or Early Termination. Subjects are eligible for enrollment if they have facial non-cystic acne with a global severity grade of a 2 (mild) or a 3 (moderate) on the Modified IGA scale at Baseline.

SECONDARY OUTCOMES:
Change in Non-Cystic Acne Quality of Life questionnaire scores | Baseline to Day 84
  The Non-Cystic Acne Quality of Life questionnaire will ask subjects a series of questions to assess the impact of this therapy on their daily quality of life in relation to their facial non-cystic acne. A decrease in response values at Day 84 indicates a change compared to baseline response values. Scale is 0 to 4.
Change in Non-Cystic Acne Self Assessment questionnaire scores | Baseline to Day 84
  The Non-Cystic Acne Self-Assessment Questionnaire will ask subjects a series of questions related to their facial non-cystic acne. A decrease in response values at Day 84 indicates a change compared to baseline response values. Scale is 0 to 4.
Change in Analysis of the Clear Skin Formula Supplement Subject Satisfaction questionnaire | Day 84/End of Study
  The Clear Skin Formula Supplement Subject Satisfaction Questionnaire will ask subjects a series of questions related to their opinion of the treatment satisfaction and ease of use at the Day 84 visit. Change in analysis at Day 84 would be indicated by low response values. Score is 1 to 5.

OTHER OUTCOMES:
Change in the VISIA photography imaging of the left, right and front views of the face to include the (1) Percentile Rating, (2) Score Rating and (3) Feature Count Rating for Wrinkles, Texture, Pores, Red Areas and Porphyrins. | Baseline to Day 84
  Subjects will have VISIA Facial imaging photographs taken of the right, central and left views of the face. All VISIA facial images will be analyzed to acquire the following data points: (1) WRINKLES - The light green lines represent fine lines and the dark green lines represent deeper wrinkles. Improvement is shown by the dark green lines turning to light green and/or the light green lines going away (2) TEXTURE- Texture is the overall smoothness of the surface of the skin, where the skin raises and dips down. The yellow dots show where the skin is raised, the blue dots show where the skin dips down. (3) PORES - Enlarged pores only (4) RED AREAS -The vascular condition, anything to do with the blood will be picked up in the reds, telangiectasia, rosacea, broken capillaries, spider veins, acne etc. (5) PORPHYRINS - This is bacteria, basically an excretion of P-acnes. Someone with oily skin will have a higher porphyrin score. Scores are 0 to 100.
The frequency of both local and systemic AEs | Baseline, Day 14, Day 28, Day 56 and Day 84 or End of Study (up to 12 weeks)
  An adverse event is any adverse change from the subject's baseline condition, i.e. any subjective signs and symptoms, or change in a concomitant disease present at the screening visit. This includes inter-current signs, symptoms, illness and significant deviations from baseline which may occur during the course of the clinical study, whether considered related to treatment or not.
Investigator Tolerability Assessment (erythema, edema, dryness, scaling, hypopigmentation and hyperpigmentation) | Baseline, Day 14, Day 28, Day 56 and Day 84 or End of Study (up to 12 weeks)
  Investigator Tolerability evaluations will be performed at Baseline, Day 14, Day 28, Day 56, Day 84 or Early Termination. Local cutaneous tolerability will be evaluated by the Investigator to assess the signs of erythema, edema, dryness, scaling, hypopigmentation and hyperpigmentation on the global facial area at Baseline and subjects will report the degree of any of these symptoms they have experienced since the previous time point. Scale is 0 to 3 with lower scores indicating a better outcome.
Subject Tolerability Self-Assessment (itching, burning and stinging) | Baseline, Day 14, Day 28, Day 56 and Day 84 or End of Study (up to 12 weeks)
  Subject Tolerability evaluations will be performed at Baseline, Day 14, Day 28, Day 56, Day 84 or Early Termination. Local cutaneous tolerability will be evaluated by the subject reporting the degree of burning, itching, and stinging on the global facial area at Baseline and subjects will report the degree of any of these symptoms they have experienced since the previous time point. Scale is 0 to 3 with lower scores indicating a better outcome.
Changes in Clinical laboratory analyses of Complete Blood Count without Differential and with Platelets | Baseline to Day 84
  Number of participants with abnormal clinical laboratory analyses of Complete Blood Count without Differential and with Platelets Panel (this is a single blood panel). The analyses will be conducted on blood samples collected from subjects at Baseline and Week 12. All results will be reported, including results that are abnormal.
  The Complete Blood Count without Differential and with Platelets Panel (single blood panel) contains the following tests:
  WBC RBC Hemoglobin Hematocrit MCV MCH MCHC RDW Platelets
Changes in Clinical laboratory analyses of Complete Metabolic Panel | Baseline to Day 84
  Number of participants with abnormal clinical laboratory analyses of Complete Metabolic Panel (this is a single blood panel). The analyses will be conducted on blood samples collected from subjects at Baseline and Week 12. All results will be reported, including results that are abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- Ablon Skin Institute & Research Center, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ablon G. A 12-week, Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of a Nutraceutical Supplement for Mild to Moderate Non-cystic Acne in Young Adults. J Clin Aesthet Dermatol. 2024 Nov;17(11):24-30. PMID 39758223